CLINICAL TRIAL: NCT06626867
Title: Effect of Dietary Fiber on Metabolic Syndrome, Gastrointestinal Function, Mood and Sleep Quality
Brief Title: Effect of Dietary Fiber on Metabolic Syndrome, Gastrointestinal Function, Mood and Sleep Quality in Obese People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chien-Wen Hou (Other)
Responsible Party: Sponsor-Investigator, Chien-Wen Hou, professor, University of Taipei
Organization: University of Taipei (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021006001
Record Dates: First submitted 2024-09-01; First posted 2024-10-04 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Hypertension; Hyperglycemia; Dyslipidemia; Obesity; Metabolic Syndrome
Keywords: prebiotic; POMS; PSQI; indigestible dextrin; dietary fiber
MeSH Terms: conditions — Hypertension; Hyperglycemia; Dyslipidemias; Obesity; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Placebo Comparator): Ingest maltodextrin
  Interventions: Other: Placebo
- dietary fiber (Experimental): Ingest indigestible dextrin supplementation
  Interventions: Dietary Supplement: Dietary Fiber Supplementation

INTERVENTIONS:
Dietary Supplement: Dietary Fiber Supplementation — Each participant ingested either dietary fiber or placebo. The dietary fiber is indi-gestible dextrin (The WiseMan's Dining, KING CAR OTSUKA CO., Taipei, Taiwan). The dosage of contents in each package is 6 grams, 3 packs a day, with a total dose of 18 grams.
  Arms: dietary fiber
Other: Placebo — The placebo was a colored capsule with 5 grams of maltodextrin, which is taken once a day.
  Arms: placebo

SUMMARY:
Metabolic syndrome includes hypertension(high blood pressure), hyperglycemia(high blood suger), dyslipidemia(abnormal blood lipid level) and obesity. The more items that meet metabolic syndrome, the higher the risk of cardiovascular disease and diabetes, and the higher the combined mortality. At present, research reports point out that the occurrence of metabolic syndrome is related to age, obesity, lifestyle and genetics.

The lack of sleep may reduce the diversity of intestinal flora, and conversely, if the diversity of intestinal flora can be increased, the quality of sleep may be improved. Dietary fiber can improve intestinal microflora and related indexes of metabolic syndrome.

Although recent studies have demonstrated that dietary fiber will affect obesity, mood and sleep, different kinds of dietary fiber will affect different strains and pro-duce different effects. The effect of resistant starch on metabolic syndrome, mood and sleep of obese people is not very clear. Therefore, the objective of this intervention trial was to evaluate the effects of the intake of resistant starch on sleep, mood, changes in body composition and biomarkers in metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Obese working popu-lation aged between 30 and 45;
* Body fat is more than 25% for male and more than 30% for female

Exclusion Criteria:

* Taking any medicines;
* Menopausal women;
* Pregnant woman

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-05-08 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Body fat percentage | From enrollment to the end of treatment at 8 weeks
  Body fat percentage was estimated by dual-energy X-ray absorptiometry (DEXA; GE Lunar Prodigy 8743, Madison, WI, USA). The same experienced technician performed the analysis of the scan.
Fasting glucose | From enrollment to the end of treatment at 8 weeks
  Fasting blood samples were obtained at morning after the participants had 12 h of overnight fasting. To obtain plasma or serum, the blood samples with 5 ml collected into blood sampling tubes with or without ethylene diamine tetraacetic acid (EDTA), respectively, were centrifuged at 3000 rpm at 4 °C for 15 min and then stored at -80 °C until analysis. The plasma blood samples were assessed using fully automated analyz-er (AU5800, Beckman Coulter®, America). A set of standard samples will be collected and analysed on the same day, including fasting glucose(mmol/L).
Mood disturbance(Questionnaires) | From enrollment to the end of treatment at 8 weeks
  The Profile of Mood States, Revised (POMS-R) is an updated version of the original Profile of Mood States (POMS) questionnaire. It is a self-report tool used to assess a person's mood by measuring different dimensions of affective states, include:
  1. Tension
  2. Depression
  3. Anger
  4. Fatigue
  5. Confusion
  6. Vigor Total Mood Disturbance (TMD) score=(Sum of negative mood scores)-Vigor score. Higher scores in the negative mood dimensions (T, D, A, F, C) indicate greater mood disturbances, while a higher score in Vigor-Activity reflects a more positive mood. The TMD score reflects overall mood disturbance, with higher TMD indicating more severe mood issues.
  This scoring system helps provide a snapshot of a person's emotional state across various mood domains.
Pittsburgh Sleep Quality Index(Questionnaires) | From enrollment to the end of treatment at 8 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire used to assess sleep quality over a 1-month period. It includes 19 items grouped into seven components:
  1. Subjective sleep quality - An individual's perception of their sleep quality.
  2. Sleep latency - The amount of time it takes to fall asleep.
  3. Sleep duration - The total amount of sleep per night.
  4. Habitual sleep efficiency - The ratio of total sleep time to time spent in bed.
  5. Sleep disturbances - The frequency of waking up due to various factors (e.g., needing to use the bathroom, feeling too hot/cold, or being disturbed by noise).
  6. Use of sleep medication - The frequency and use of medication to help sleep.
  7. Daytime dysfunction - Difficulties staying awake during the day or performing daily activities due to poor sleep.
  Each component is scored from 0 to 3, with a total score range of 0 to 21. A score above 5 indicates poor sleep quality.
Biochemical Markers | From enrollment to the end of treatment at 8 weeks
  Fasting blood samples were obtained at morning after the participants had 12 h of overnight fasting. To obtain plasma or serum, the blood samples with 5 ml collected into blood sampling tubes with or without ethylene diamine tetraacetic acid (EDTA), respectively, were centrifuged at 3000 rpm at 4 °C for 15 min and then stored at -80 °C until analysis. The plasma blood samples were assessed using fully automated analyz-er (AU5800, Beckman Coulter®, America). A set of standard samples will be collected and analysed on the same day, including fasting glucose, high sensitivity C-reactive protein (HsCRP), fasting insulin, total cholesterol, low density lipoprotein (LDL-C), high density lipoprotein (HDL-C) and triglyceride (TG). Insulin was measured by us-ing electrochemiluminescence immunoassay (ECLIA) (Cobas e801, Roche Diagnostics, Mannheim, Germany); glycated hemoglobin (HbA1c) was measured by using an ion exchange resin composed of hydrophilic polymer of methacrylate ester copolymer (H
High sensitivity C-reactive protein | From enrollment to the end of treatment at 8 weeks
  Fasting blood samples were obtained at morning after the participants had 12 h of overnight fasting. To obtain plasma or serum, the blood samples with 5 ml collected into blood sampling tubes with or without ethylene diamine tetraacetic acid (EDTA), respectively, were centrifuged at 3000 rpm at 4 °C for 15 min and then stored at -80 °C until analysis. The plasma blood samples were assessed using fully automated analyz-er (AU5800, Beckman Coulter®, America). A set of standard samples will be collected and analysed on the same day, including high sensitivity C-reactive protein (HsCRP)(mg/L).
Total cholesterol | From enrollment to the end of treatment at 8 weeks
  Fasting blood samples were obtained at morning after the participants had 12 h of overnight fasting. To obtain plasma or serum, the blood samples with 5 ml collected into blood sampling tubes with or without ethylene diamine tetraacetic acid (EDTA), respectively, were centrifuged at 3000 rpm at 4 °C for 15 min and then stored at -80 °C until analysis. The plasma blood samples were assessed using fully automated analyz-er (AU5800, Beckman Coulter®, America). A set of standard samples will be collected and analysed on the same day, including total cholesterol(mmol/L).
Triglyceride | From enrollment to the end of treatment at 8 weeks
  Fasting blood samples were obtained at morning after the participants had 12 h of overnight fasting. To obtain plasma or serum, the blood samples with 5 ml collected into blood sampling tubes with or without ethylene diamine tetraacetic acid (EDTA), respectively, were centrifuged at 3000 rpm at 4 °C for 15 min and then stored at -80 °C until analysis. The plasma blood samples were assessed using fully automated analyz-er (AU5800, Beckman Coulter®, America). A set of standard samples will be collected and analysed on the same day, including triglyceride (TG)(mmol/L).

SECONDARY OUTCOMES:
Blood pressure | From enrollment to the end of treatment at 8 weeks
  Blood pressure will be measured from the non-dominant arm with a digital blood pressure monitor (Omron HEM-7121, Japan) in sitting position after at least 15 min of rest, including diastolic blood pressure and systolic blood pressure.
Anthropometrics | From enrollment to the end of treatment at 8 weeks
  Body height and weight will be measured on a stadiometer (Takei Scientific In-struments, Tokyo, Japan) and digital scale (TANITA WB-110MA, Tokyo, Japan) to the nearest 0.1 cm and 0.1 kg without shoes and wearing light clothes. Waist circumference was measured at the midpoint between the iliac crest and the lowest rib margin, and hip circumference was assessed at the widest point around the buttocks. Based on the anthropometric metric measures, body mass index (BMI; kg/m2) and waist to hip ratio (WHR; waist/hip) were calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Exercise Biochemistry, Department of Sports Sciences, University of Taipei, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No